CLINICAL TRIAL: NCT04759677
Title: Energy Expenditure And Exercise Intensity Of Interactive Video Gaming in Cerebral Palsy: Hip Versus Wrist Accelerometer Data
Brief Title: Exercise Intensity Of Interactive Video Gaming in Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Pınar Ciddi, Assistant Orofessor, Medipol University
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: E-10840098-772.02-2683
Record Dates: First submitted 2021-02-10; First posted 2021-02-18 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: Cerebral Palsy
Keywords: energy expenditure; exercise intensity; video games
MeSH Terms: conditions — Cerebral Palsy | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: All 20 individuals with CP will participate in a total of 2 exercise sessions on consecutive days with 45 minutes of active video games. During the training sessions, exercise intensity will be evaluated with the accelerometer.
  The accelerometer will be placed on the dominant wrist of 20 individuals during one training session. The same 20 individuals will participate in the other exercise session and the accelerometer will be placed on the dominant side hip area of the individuals this time. Exercise intensity values obtained from 2 different training sessions will be compared.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the situation where the accelerometer is placed on the wrist during active video games playing (Active Comparator): In one session the accelerometer will place on the dominant wrist Individuals will instructed not to remove and instruct them to wear the device during the session.
  Interventions: Other: Exercise with active video games
- the situation where the accelerometer is placed on the hip during active video games playing (Active Comparator): In one session the accelerometer will place on a flexible belt by attaching to the hip area at the intersection of the dominant wrist and axillary line.
  Individuals will instructed not to remove and instruct them to wear the device during the session.
  Interventions: Other: Exercise with active video games

INTERVENTIONS:
Other: Exercise with active video games — 45-minute exercise in which individuals played pre-selected games from Nintendo Wii while keeping in mind their functional level, skills and needs. Four Nintendo Wii games were chosen: Island Cycling, Tilt Table Balance Board, Soccer Heading and Boxing. Each and every individual played these given four games consecutively in one session.

SUMMARY:
The purpose of this study is to compare the energy consumption and exercise intensities obtained from an activity classifier obtained from a triaxial acceleration signal collected from the wrist and hip during active video games in children with ambulated Cerebral Palsy. .

All 20 individuals with CP will participate in a total of 2 exercise sessions on consecutive days with 45 minutes of active video games. In two exercise season individuals will play 4 games that were previously determined and experienced for about 45 minutes. During the training sessions, exercise intensity will be evaluated with the accelerometer.

The accelerometer will be placed on the dominant wrist of 20 individuals during one training session. The same 20 individuals will participate in the other exercise session and the accelerometer will be placed on the dominant side hip area of the individuals this time. Exercise intensity values obtained from 2 different training sessions will be compared.

Exercise intensity will be measured by an ActiGraph wGT3X-BT triaxial accelerometer during the interventions.

For both intervention sessions, a statistical comparison will made between groups in terms of energy consumption, activity counts, and active duration.

DETAILED DESCRIPTION:
More validation studies are needed to document the most appropriate place (wrist or waist) to capture limb movement and / or energy consumption (capturing) during physical activity in children with CP at different functional levels. Such information has the potential to guide interventions to improve daily activity throughout life, with potential implications for participation and quality of life.

The purpose of this study is to compare the energy consumption and exercise intensities obtained from an activity classifier obtained from a triaxial acceleration signal collected from the wrist and hip during active video games in children with ambulated Cerebral Palsy. Thus, it is thought that reaching the targeted physical activity intensity with active video games in individuals with CP in the clinic can be evaluated with an appropriate and accurate accelerometer placement.

Functional levels of individuals will be determined according to GMFCS. All 20 individuals with CP will participate in a total of 2 exercise sessions with on consecutive days with 45 minutes of active video games. In two exercise season individuals will play 4 games that were previously determined and experienced for about 45 minutes. During the training sessions, exercise intensity will be evaluated with the accelerometer.

The accelerometer will be placed on the dominant wrist of 20 individuals during one training session. The same 20 individuals will participate in the other exercise session and the accelerometer will be placed on the dominant side hip area of the individuals this time. Exercise intensity values obtained from 2 different training sessions will be compared.

Exercise intensity (energy consumption (MET), activity counts, active time during session) will be measured by an ActiGraph wGT3X-BT triaxial accelerometer during the interventions. After the measurements were over, the accelerometer data will be loaded on a personal computer and manipulated in ActiLife software version 6.13.3.

For both intervention sessions, a statistical comparison will made between groups in terms of energy consumption, activity counts, and active duration. Statistical analysis will be performed using SPSSc 22.00 package program. Number and percentage will be used for demographic data, mean ± standard deviation notation and descriptive data. In the dependent variables, inter-measurement changes will be evaluated with Wilcoxon test, inter-measurement changes in independent variables will be evaluated by Mann Whitney U test.

ELIGIBILITY:
Inclusion Criteria

* must be at I-III level according to the Gross Motor Function Classification System (GMFCS)
* must be able to cooperate during assessments and exercise sessions
* must have sufficient functional dexterity to grasp the Nintendo Wii remote control

Exclusion Criteria:

* having excessive upper extremity spasticity that can interfere with movements while playing
* playing Nintendo Wii before
* genetic or neurological disease other than CP diagnosis and epilepsy
* having had muscle-tendon and bone surgery less than 6 months ago
* use of any pharmacological agent to inhibit spasticity less than 6 months ago

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Energy consumption (MET) Exercise Intensity | up to 2 days
  Energy consumption will be measured by an ActiGraph wGT3X-BT triaxial accelerometer during the exercise sessions
Activity counts | up to 2 days
  Activity counts will be measured by an ActiGraph wGT3X-BT triaxial accelerometer during the exercise sessions
Active time | up to 2 days
  Active time will be measured by an ActiGraph wGT3X-BT triaxial accelerometer during the exercise sessions

CONTACTS AND LOCATIONS:
Overall Officials: Pınar Kaya Ciddi, Principal Investigator — İstanbul Medipol University
Locations (1):
- Medipol University, Istanbul, Beykoz, Turkey (Türkiye)